CLINICAL TRIAL: NCT04205643
Title: A Randomized, Placebo Controlled, Double-Blind, Phase 3 Study to Evaluate the Efficacy and Safety of the Subcutaneous Injection of CT-P13 (CT-P13 SC) as Maintenance Therapy in Patients With Moderately to Severely Active Ulcerative Colitis
Brief Title: CT-P13 (Infliximab) Subcutaneous Administration in Patients With Moderately to Severely Active Ulcerative Colitis (LIBERTY-UC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P13 3.7; 2019-003849-15 (EudraCT Number)
Record Dates: First submitted 2019-12-18; First posted 2019-12-19 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-08

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CT-P13 SC (Experimental)
  Interventions: Biological: CT-P13 SC (Infliximab)
- Placebo SC (Placebo Comparator)
  Interventions: Other: Placebo SC

INTERVENTIONS:
Biological: CT-P13 SC (Infliximab) — Subcutaneous injection of CT-P13 SC
  Arms: CT-P13 SC
Other: Placebo SC — Subcutaneous injection of Placebo SC
  Arms: Placebo SC

SUMMARY:
This is Phase 3, Randomized, Placebo-controlled study to demonstrate superiority of CT-P13 SC over Placebo SC in Patients With Moderately to Severely Active Ulcerative Colitis

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female aged 18 to 75 years, inclusive.
* Patient has moderately to severely active UC with a modified Mayo score of 5 to 9 points with endoscopic subscore of ≥ 2 points

Exclusion Criteria:

* Patient who has previously received 2 or more biologic agents and/or JAK inhibitors
* Patient who has previously received either a TNFα inhibitor or biologic agent within 5 half-lives

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 548 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2023-07-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centrum Zdrowia MDM, Warsaw, Poland

REFERENCES:
- [Derived] Colombel JF, Sandborn WJ, Schreiber S, Danese S, Klopocka M, Kierkus J, Kulynych R, Gonciarz M, Soltysiak A, Smolinski P, Sreckovic S, Valuyskikh E, Lahat A, Horynski M, Gasbarrini A, Osipenko M, Borzan V, Kowalski M, Saenko D, Sardinov R, Lee SJ, Kim S, Bae Y, Lee S, Lee S, Lee JH, Kim JM, Park G, Lee J, Lee J, Ryu JY, Sands BE, Hanauer SB. Subcutaneous infliximab (CT-P13 SC) as maintenance therapy for Crohn's disease and ulcerative colitis: 2-year results from open-label extensions of two randomized controlled trials (LIBERTY). J Crohns Colitis. 2025 Jun 4;19(6):jjaf060. doi: 10.1093/ecco-jcc/jjaf060. PMID 40243842
- [Derived] Hanauer SB, Sands BE, Schreiber S, Danese S, Klopocka M, Kierkus J, Kulynych R, Gonciarz M, Soltysiak A, Smolinski P, Sreckovic S, Valuyskikh E, Lahat A, Horynski M, Gasbarrini A, Osipenko M, Borzan V, Kowalski M, Saenko D, Sardinov R, Lee SJ, Kim S, Bae Y, Lee S, Lee S, Lee JH, Yang S, Lee J, Lee J, Kim JM, Park G, Sandborn WJ, Colombel JF. Subcutaneous Infliximab (CT-P13 SC) as Maintenance Therapy for Inflammatory Bowel Disease: Two Randomized Phase 3 Trials (LIBERTY). Gastroenterology. 2024 Oct;167(5):919-933. doi: 10.1053/j.gastro.2024.05.006. Epub 2024 May 23. PMID 38788861

RESULTS

PARTICIPANT FLOW:
Groups:
- CT-P13 IV 5mg/kg: Induction phase: Patients who enrolled received induction doses of CT-P13 5mg/kg via intravenous (IV) infusion at Weeks 0, 2, and 6.
- CT-P13 SC 120 mg: Maintenance phase: Patients who were classified as clinical responder at Week 10 received CT-P13 120mg subcutaneously every 2 weeks from Week 10 to Week 54.
  From Week 22, patients who initially responded but then lost response could increase the dose to CT-P13 SC 240mg (double injection [2 shots] of CT-P13 SC 120 mg) every 2 weeks.
- Placebo: Maintenance phase: Patients who were classified as clinical responder at Week 10 received placebo-matching subcutaneously every 2 weeks from Week 10 to Week 54.
  From Week 22, patients who initially responded but then lost response could increase the dose to CT-P13 SC 240mg (double injection [2 shots] of CT-P13 SC 120 mg) every 2 weeks.
Period: Induction Phase
Arm/Group | CT-P13 IV 5mg/kg | CT-P13 SC 120 mg | Placebo
Started | 548 | 0 | 0
Completed | 438 | 0 | 0
Not Completed | 110 | 0 | 0
Period: Maintenance Phase
Arm/Group | CT-P13 IV 5mg/kg | CT-P13 SC 120 mg | Placebo
Started | 0 | 294 | 144
Completed | 0 | 240 | 113
Not Completed | 0 | 54 | 31

BASELINE CHARACTERISTICS:
Population: All-randomized population
Groups:
- CT-P13 SC 120 mg: CT-P13 SC 120 mg
- Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | CT-P13 SC 120 mg | Placebo | Total
Number analyzed (Participants) | 294 | 144 | 438
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (12.78) | 40.4 (13.49) | 38.9 (13.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 131 | 61 | 192
  Male | 163 | 83 | 246
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 4 | 10
  White | 288 | 140 | 428
Region of Enrollment [Number; unit: participants]
  Belarus | 3 | 0 | 3
  Bulgaria | 4 | 2 | 6
  Croatia | 9 | 2 | 11
  Czechia | 5 | 6 | 11
  Israel | 2 | 1 | 3
  Italy | 10 | 5 | 15
  Latvia | 3 | 1 | 4
  Mexico | 6 | 4 | 10
  Poland | 135 | 65 | 200
  Russia | 56 | 21 | 77
  Serbia | 12 | 8 | 20
  South Africa | 2 | 1 | 3
  Turkey | 7 | 2 | 9
  Ukraine | 40 | 26 | 66

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving Clinical Remission at Week 54
Description: Clinical remission defined by modified Mayo score which ranges from 0 to 9, including Stool frequency subscore, Rectal bleeding subscore and Endoscopic subscore but excluding Physician's global assessment subscore from the Total Mayo score.
  Patients with dose adjustment to CT-P13 SC 240 mg prior to Week 54 were considered as non-remitter.
Time Frame: Week 54
Population: All-randomized population
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 SC 120 mg | Placebo
Number analyzed (Participants) | 294 | 144
Participants | 127 | 30
Statistical Analysis 1: Comparison: CT-P13 SC 120 mg; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — If the primary endpoint is significant, a fixed sequence procedure was employed to control the overall type I error rate of the key secondary endpoints; Stratified by Previous biologic agent and/or JAK inhibitors exposure, Use of oral corticosteroids treatment at Week 0, Clinical remission at Week 10; Difference estimated using CMH weights = 21.1, 95% CI 2-sided [11.8 to 29.3] — The 95% stratified Newcombe CI with CMH weights

2. Secondary Outcome: Percentage Patients Achieving Clinical Response at Week 54
Description: Clinical response defined by decrease in modified Mayo score from baseline of at least 2 points and at least 30%, with an accompanying decrease in the rectal bleeding subscore of at least 1 point or an absolute rectal bleeding subscore of 0 or 1 point. Patients with dose adjustment to CT-P13 SC 240 mg prior to Week 54 were considered as non-responder.
Time Frame: Week 54
Population: All-randomized population
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 SC 120 mg | Placebo
Number analyzed (Participants) | 294 | 144
Participants | 158 | 45

3. Secondary Outcome: Percentage of Patients Achieving Endoscopic-Histologic Mucosal Improvement at Week 54
Description: Endoscopic-histologic mucosal improvement defined as an absolute endoscopic subscore of 0 or 1 point from modified Mayo score and an absolute RHI score of 3 points or less with an accompanying lamina propria neutrophils and neutrophils in epithelium subscore of 0 point. Patients with dose adjustment to CT-P13 SC 240 mg prior to Week 54 were considered as endoscopic-histologic mucosal improvement not achieved.
Time Frame: Week 54
Population: All-randomized population
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 SC 120 mg | Placebo
Number analyzed (Participants) | 294 | 144
Participants | 105 | 24

4. Secondary Outcome: Percentage of Patients Achieving Corticosteroid-Free Remission at Week 54
Description: Corticosteroid-free remission defined as being in clinical remission by modified Mayo score in addition to not requiring any treatment with corticosteroid for at least 8 weeks at Week 54, among the patients who used oral corticosteroids at baseline. Patients with dose adjustment to CT-P13 SC 240 mg prior to Week 54 were considered as non-remitter.
Time Frame: Week 54
Population: Patients who used oral corticosteroids at baseline among the All-randomized population
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P13 SC 120 mg | Placebo
Number analyzed (Participants) | 120 | 61
Participants | 44 | 11

ADVERSE EVENTS:
Time Frame: For CT-P13 SC and Placebo groups, the overall summary of Treatment-Emergent Adverse Events during the maintenance period (from Week 10 to Week 54) was reported. For CT-P13 IV 5mg/kg group, the overall summary of Treatment-Emergent Adverse Events during the induction phase (from Week 0 to prior to Week 10, before initiation of CT-P13 SC administeration) was reported.
Description: Safety analyses were pre-specified to only report the most severe event if the same events were occurred to the same patient.
  For CT-P13 IV 5mg/kg group, the safety analyses were performed ITT population. For CT-P13 SC and Placebo groups, the safety analyses were performed in the safety population. Analysis of safety population were performed based on the actual treatment group and differences from the randomized population accordingly.
Groups:
- CT-P13 IV 5 mg/kg: Patients who administered CT-P13 IV 5mg/kg at Week 0, 2, and 6.
- CT-P13 SC 120 mg: Patients who administered CT-P13 SC 120 mg every 2 weeks from W10 to Week 54. Patients who received adjusted dose of CT-P13 SC 240mg which is allowed from Week 22 are also included.
- Placebo: Patients who administered Placebo every 2 weeks from W10 to Week 54. For patients who received adjusted dose of CT-P13 SC 240mg, data collected before initiation of dose adjustment are included.
Arm/Group | CT-P13 IV 5 mg/kg | CT-P13 SC 120 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/548 | 0/296 | 0/140
Serious Adverse Events (participants affected / at risk) | 23/548 | 15/296 | 4/140
Other Adverse Events (participants affected / at risk) | 89/548 | 60/296 | 37/140
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P13 IV 5 mg/kg (N=548) | CT-P13 SC 120 mg (N=296) | Placebo (N=140)
Anaemia (Study drug unrelated) (Blood and lymphatic system disorders) | 3 | 1 | 0
Iron deficiency anaemia (study drug unrelated) (Blood and lymphatic system disorders) | 2 | 1 | 0
Aortic valve incompetence (study drug unrelated) (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (study drug unrelated) (Cardiac disorders) | 0 | 1 | 0
Colitis ulcerative (study drug unrelated) (Gastrointestinal disorders) | 3 | 2 | 1
Duodenal ulcer (study drug unrelated) (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer perforation (study drug unrelated) (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (study drug unrelated) (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal strangulation (study drug unrelated) (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine perforation (study drug unrelated) (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis acute (study drug related) (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (study drug unrelated) (Gastrointestinal disorders) | 0 | 0 | 1
Appendicitis (study drug unrelated) (Infections and infestations) | 1 | 0 | 0
COVID-19 (study drug unrelated) (Infections and infestations) | 1 | 1 | 0
COVID-19 pneumonia (study drug unrelated) (Infections and infestations) | 2 | 2 | 0
Cellulitis (study drug related) (Infections and infestations) | 1 | 0 | 1
Cystitis (study drug unrelated) (Infections and infestations) | 0 | 1 | 0
Cytomegalovirus infection (study drug unrelated) (Infections and infestations) | 2 | 0 | 0
Peritonitis (study drug unrelated) (Infections and infestations) | 1 | 0 | 0
Pneumonia (study drug related) (Infections and infestations) | 0 | 1 | 0
Salpingitis (study drug unrelated) (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (study drug related) (Infections and infestations) | 0 | 1 | 0
Urosepsis (study drug unrelated) (Infections and infestations) | 1 | 0 | 0
Anastomic leak (study drug unrelated) (Injury, poisoning and procedural complications) | 1 | 0 | 0
Clavicle fracture (study drug unrelated) (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (study drug related) (Injury, poisoning and procedural complications) | 3 | 0 | 0
Arthritis (study drug unrelated) (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Colorectal adenoma (study drug unrelated) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neuromyopathy (study drug unrelated) (Nervous system disorders) | 0 | 0 | 1
Ureterolithiasis (study drug unrelated) (Renal and urinary disorders) | 1 | 0 | 0
Cervical dysplasia (study drug unrelated) (Reproductive system and breast disorders) | 1 | 0 | 0
Deep vein thrombosis (study drug unrelated) (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P13 IV 5 mg/kg (N=548) | CT-P13 SC 120 mg (N=296) | Placebo (N=140)
Anaemia (Blood and lymphatic system disorders) | 34 | 11 | 5
Colitis ulcerative (Gastrointestinal disorders) | 13 | 13 | 13
COVID-19 (Infections and infestations) | 13 | 26 | 9
Nasopharyngitis (Infections and infestations) | 9 | 5 | 7
Headache (Nervous system disorders) | 30 | 15 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT04205643/Prot_002.pdf
  • Statistical Analysis Plan (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT04205643/SAP_001.pdf